CLINICAL TRIAL: NCT03018236
Title: The Effect of N-acetylcysteine (NAC) on Treatment of Alcohol and Cocaine Use Disorders: A Double-Blind Randomized Controlled Trial.
Brief Title: Effect of N-acetylcysteine on Alcohol and Cocaine Use Disorders: A Double-Blind Randomized Controlled Trial.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Secretaria Nacional de Políticas sobre Drogas (SENAD) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 150488
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Cocaine Addiction; Alcohol Addiction
Keywords: cocaine; alcohol; substance use disorders; addiction; N-acetylcysteine; randomized controlled trial
MeSH Terms: conditions — Cocaine-Related Disorders; Alcoholism; Substance-Related Disorders; Behavior, Addictive | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Alcohol N-acetylcysteine (Experimental): 600 mg N-acetylcysteine capsule by mouth, every 12 hours for 8 weeks
  Interventions: Drug: Alcohol N-acetylcysteine
- Alcohol Placebo (Placebo Comparator): A placebo capsule matching color and smell of the active medication
  Interventions: Drug: Alcohol Placebo
- Cocaine N-acetylcysteine (Experimental): 600 mg N-acetylcysteine capsule by mouth, every 12 hours for 8 weeks
  Interventions: Drug: Cocaine N-acetylcysteine
- Cocaine Placebo (Placebo Comparator): A placebo capsule matching color and smell of the active medication
  Interventions: Drug: Cocaine Placebo

INTERVENTIONS:
Drug: Alcohol N-acetylcysteine — 1200 mg of NAC per day, taken in two doses, for subjects with alcohol use disorder
  Other Names: NAC
  Arms: Alcohol N-acetylcysteine
Drug: Alcohol Placebo — Flour pills looking exactly the same as the active compound, for subjects with alcohol use disorder
  Arms: Alcohol Placebo
Drug: Cocaine N-acetylcysteine — 1200 mg of NAC per day, taken in two doses, for subjects with cocaine use disorder
  Other Names: NAC
  Arms: Cocaine N-acetylcysteine
Drug: Cocaine Placebo — Flour pills looking exactly the same as the active compound, for subjects with cocaine use disorder
  Arms: Cocaine Placebo

SUMMARY:
This study evaluates the use of N-acetylcysteine in the treatment of alcohol and cocaine use disorders. Alcohol users will be split in two groups, one will receive the active N-acetylcysteine and the other placebo. The same division will occur with cocaine users. The effects of N-acetylcysteine in adherence, abstinence, psychiatric symptoms and stress biomarkers will be evaluated.

DETAILED DESCRIPTION:
N-acetylcysteine acts replenishing the human body glutathione storages. Glutathione is an important antioxidant agent, and also modulates the N-methyl-D-aspartate (NMDA) glutamatergic receptor. Glutamate has been associated with the neuroadaptation related to substance use disorders, and thus it is considered a potential target for pharmacological interventions regarding these disorders. N-acetylcysteine also interacts with the cystine-glutamate antiporter on astrocytes hence increasing glutamate release into the extracellular space.

N-acetylcysteine effects and its implications in the addiction disorders have been studied initially with animal models. Glutamate levels normalization through N-acetylcysteine reduced compulsive drug self-administration and drug-seeking behavior in mice. In addition, there are promising results also with human subjects, showing benefits for cocaine, alcohol and cannabis use disorders.

This study consists of a randomized, double-blind, placebo controlled trial with four arms: alcohol users divided into NAC vs Placebo and cocaine users divided into NAC vs Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of Alcohol or Cocaine Use Disorder
* Seven days of inpatient treatment in an addiction treatment specialized unit

Exclusion Criteria:

* Another Substance Use Disorder (exception: tobacco)
* Severe medical conditions (cardiac, renal or hepatic), that preclude subject participation
* History of asthma or convulsions medication use
* Recent use (<14 days) of any medication that could interfere with the study medication
* History of anaphylactic reactions with the study medication
* Suicide risk
* Inability to understand the informed consent form or to comply with the study requirements
* Any severe neuropsychiatric condition, not caused by the substance use, that requires specific medication treatments and could interfere with the study development, in the investigators opinion (for instance: dementia, schizophrenia or other psychoses, multiple sclerosis, severe depression, stroke, epilepsy, bipolar disorder)
* Failing to complete the screening procedures prior to the study first week

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants who attended all study appointments | 8 weeks
  Completers (i.e. subjects who attended all study appointments) vs non-completers

SECONDARY OUTCOMES:
Abstinence by urine | 8 weeks
  Amount of positive urine tests for cocaine users
Abstinence by breathalyzer | 8 weeks
  Amount of positive breathalyzer tests for alcohol users
Abstinence by self report | 8 weeks
  Timeline Followback Method
Days of inpatient treatment | Up to 4 weeks
  The difference (if any) between placebo and intervention groups in the amount of inpatient treatment days.
Change in scores of CGI | 8 weeks
  Differences in scores of the Clinical Global Impression (CGI)
Change in scores of FAST | 8 weeks
  Differences in scores of the Functioning Assessment Short Test (FAST).
Depressive symptoms | 8 weeks
  Differences in scores of the Beck Depression Inventory (BDI)
Anxiety symptoms | 8 weeks
  Differences in scores of the Beck Anxiety Inventory (BAI)
BDNF | 8 weeks
  Differences between groups regarding dosage of Brain Derived Neurotrophic Factor (BDNF)
GSSG | 8 weeks
  Differences between groups regarding dosage of Oxidized Glutathione (GSSG)
GSH | 8 weeks
  Differences between groups regarding dosage of Glutathione (GSH)
GPx | 8 weeks
  Differences between groups regarding dosage of Glutathione Peroxidase (GPx)
CAT | 8 weeks
  Differences between groups regarding dosage of Catalase (CAT)
TBARS | 8 weeks
  Differences between groups regarding dosage of Thiobarbituric Acid Reactive Substances (TBARS)
SOD | 8 weeks
  Differences between groups regarding dosage of Superoxide Dismutase (SOD)
Carbonyl | 8 weeks
  Differences between groups regarding dosage of Carbonyl

OTHER OUTCOMES:
Adverse events | 8 weeks
  Systematic Assessment for Treatment Emergent Events (SAFTEE) application

CONTACTS AND LOCATIONS:
Overall Officials: Lisia von Diemen, PhD, Study Chair — Federal University of Rio Grande do Sul (UFRGS); Flavio Pechansky, PhD, Principal Investigator — Federal University of Rio Grande do Sul (UFRGS)
Locations (1):
- Hospital de Clinicas de Porto Alegre - Unidade Alvaro Alvim, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agrawal A, Verweij KJ, Gillespie NA, Heath AC, Lessov-Schlaggar CN, Martin NG, Nelson EC, Slutske WS, Whitfield JB, Lynskey MT. The genetics of addiction-a translational perspective. Transl Psychiatry. 2012 Jul 17;2(7):e140. doi: 10.1038/tp.2012.54. PMID 22806211
- [Background] Andreazza AC, Frey BN, Valvassori SS, Zanotto C, Gomes KM, Comim CM, Cassini C, Stertz L, Ribeiro LC, Quevedo J, Kapczinski F, Berk M, Goncalves CA. DNA damage in rats after treatment with methylphenidate. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Aug 15;31(6):1282-8. doi: 10.1016/j.pnpbp.2007.05.012. Epub 2007 Jun 2. PMID 17614179
- [Background] Baan R, Straif K, Grosse Y, Secretan B, El Ghissassi F, Bouvard V, Altieri A, Cogliano V; WHO International Agency for Research on Cancer Monograph Working Group. Carcinogenicity of alcoholic beverages. Lancet Oncol. 2007 Apr;8(4):292-3. doi: 10.1016/s1470-2045(07)70099-2. No abstract available. PMID 17431955
- [Background] Baker DA, McFarland K, Lake RW, Shen H, Toda S, Kalivas PW. N-acetyl cysteine-induced blockade of cocaine-induced reinstatement. Ann N Y Acad Sci. 2003 Nov;1003:349-51. doi: 10.1196/annals.1300.023. No abstract available. PMID 14684458
- [Background] Berk M, Malhi GS, Gray LJ, Dean OM. The promise of N-acetylcysteine in neuropsychiatry. Trends Pharmacol Sci. 2013 Mar;34(3):167-77. doi: 10.1016/j.tips.2013.01.001. Epub 2013 Jan 29. PMID 23369637
- [Background] Bibel M, Barde YA. Neurotrophins: key regulators of cell fate and cell shape in the vertebrate nervous system. Genes Dev. 2000 Dec 1;14(23):2919-37. doi: 10.1101/gad.841400. No abstract available. PMID 11114882
- [Background] Calado RT, Young NS. Telomere diseases. N Engl J Med. 2009 Dec 10;361(24):2353-65. doi: 10.1056/NEJMra0903373. No abstract available. PMID 20007561
- [Background] Chen CH, Pan CH, Chen CC, Huang MC. Increased oxidative DNA damage in patients with alcohol dependence and its correlation with alcohol withdrawal severity. Alcohol Clin Exp Res. 2011 Feb;35(2):338-44. doi: 10.1111/j.1530-0277.2010.01349.x. Epub 2010 Nov 10. PMID 21070251
- [Background] Corominas-Roso M, Roncero C, Daigre C, Grau-Lopez L, Ros-Cucurull E, Rodriguez-Cintas L, Sanchez-Mora C, Lopez MV, Ribases M, Casas M. Changes in brain-derived neurotrophic factor (BDNF) during abstinence could be associated with relapse in cocaine-dependent patients. Psychiatry Res. 2015 Feb 28;225(3):309-14. doi: 10.1016/j.psychres.2014.12.019. Epub 2014 Dec 20. PMID 25592977
- [Background] Costa MA, Girard M, Dalmay F, Malauzat D. Brain-derived neurotrophic factor serum levels in alcohol-dependent subjects 6 months after alcohol withdrawal. Alcohol Clin Exp Res. 2011 Nov;35(11):1966-73. doi: 10.1111/j.1530-0277.2011.01548.x. Epub 2011 Aug 16. PMID 21848960
- [Background] Cross CE, Valacchi G, Schock B, Wilson M, Weber S, Eiserich J, van der Vliet A. Environmental oxidant pollutant effects on biologic systems: a focus on micronutrient antioxidant-oxidant interactions. Am J Respir Crit Care Med. 2002 Dec 15;166(12 Pt 2):S44-50. doi: 10.1164/rccm.2206015. PMID 12471088
- [Background] Davis MI. Ethanol-BDNF interactions: still more questions than answers. Pharmacol Ther. 2008 Apr;118(1):36-57. doi: 10.1016/j.pharmthera.2008.01.003. Epub 2008 Feb 2. PMID 18394710
- [Background] Dean O, Giorlando F, Berk M. N-acetylcysteine in psychiatry: current therapeutic evidence and potential mechanisms of action. J Psychiatry Neurosci. 2011 Mar;36(2):78-86. doi: 10.1503/jpn.100057. PMID 21118657
- [Background] Degenhardt L, Singleton J, Calabria B, McLaren J, Kerr T, Mehta S, Kirk G, Hall WD. Mortality among cocaine users: a systematic review of cohort studies. Drug Alcohol Depend. 2011 Jan 15;113(2-3):88-95. doi: 10.1016/j.drugalcdep.2010.07.026. Epub 2010 Sep 15. PMID 20828942
- [Background] Ersche KD, Jones PS, Williams GB, Robbins TW, Bullmore ET. Cocaine dependence: a fast-track for brain ageing? Mol Psychiatry. 2013 Feb;18(2):134-5. doi: 10.1038/mp.2012.31. Epub 2012 Apr 24. No abstract available. PMID 22525488
- [Background] Frey BN, Valvassori SS, Gomes KM, Martins MR, Dal-Pizzol F, Kapczinski F, Quevedo J. Increased oxidative stress in submitochondrial particles after chronic amphetamine exposure. Brain Res. 2006 Jun 30;1097(1):224-9. doi: 10.1016/j.brainres.2006.04.076. Epub 2006 May 30. PMID 16730669
- [Background] Garbutt JC, Greenblatt AM, West SL, Morgan LC, Kampov-Polevoy A, Jordan HS, Bobashev GV. Clinical and biological moderators of response to naltrexone in alcohol dependence: a systematic review of the evidence. Addiction. 2014 Aug;109(8):1274-84. doi: 10.1111/add.12557. Epub 2014 May 23. PMID 24661324
- [Background] Grant JE, Odlaug BL, Kim SW. A double-blind, placebo-controlled study of N-acetyl cysteine plus naltrexone for methamphetamine dependence. Eur Neuropsychopharmacol. 2010 Nov;20(11):823-8. doi: 10.1016/j.euroneuro.2010.06.018. Epub 2010 Jul 22. PMID 20655182
- [Background] Gray KM, Carpenter MJ, Baker NL, DeSantis SM, Kryway E, Hartwell KJ, McRae-Clark AL, Brady KT. A double-blind randomized controlled trial of N-acetylcysteine in cannabis-dependent adolescents. Am J Psychiatry. 2012 Aug;169(8):805-12. doi: 10.1176/appi.ajp.2012.12010055. PMID 22706327
- [Background] Gray KM, Watson NL, Carpenter MJ, Larowe SD. N-acetylcysteine (NAC) in young marijuana users: an open-label pilot study. Am J Addict. 2010 Mar-Apr;19(2):187-9. doi: 10.1111/j.1521-0391.2009.00027.x. No abstract available. PMID 20163391
- [Background] Griffith JD, Rowan-Szal GA, Roark RR, Simpson DD. Contingency management in outpatient methadone treatment: a meta-analysis. Drug Alcohol Depend. 2000 Feb 1;58(1-2):55-66. doi: 10.1016/s0376-8716(99)00068-x. PMID 10669055
- [Background] Haile CN, Kosten TR, Kosten TA. Genetics of dopamine and its contribution to cocaine addiction. Behav Genet. 2007 Jan;37(1):119-45. doi: 10.1007/s10519-006-9115-2. Epub 2006 Oct 25. PMID 17063402
- [Background] Huang MC, Chen CC, Peng FC, Tang SH, Chen CH. The correlation between early alcohol withdrawal severity and oxidative stress in patients with alcohol dependence. Prog Neuropsychopharmacol Biol Psychiatry. 2009 Feb 1;33(1):66-9. doi: 10.1016/j.pnpbp.2008.10.009. Epub 2008 Oct 27. PMID 18996163
- [Background] Huang MC, Chen CH, Liu HC, Chen CC, Ho CC, Leu SJ. Differential patterns of serum brain-derived neurotrophic factor levels in alcoholic patients with and without delirium tremens during acute withdrawal. Alcohol Clin Exp Res. 2011 Jan;35(1):126-31. doi: 10.1111/j.1530-0277.2010.01329.x. Epub 2010 Oct 6. PMID 21039634
- [Background] Huang MC, Chen CH, Chen CH, Liu SC, Ho CJ, Shen WW, Leu SJ. Alterations of serum brain-derived neurotrophic factor levels in early alcohol withdrawal. Alcohol Alcohol. 2008 May-Jun;43(3):241-5. doi: 10.1093/alcalc/agm172. Epub 2008 Mar 7. PMID 18326550
- [Background] Jaffe JH. Trivializing dependence. Br J Addict. 1990 Nov;85(11):1425-7; discussion 1429-31. doi: 10.1111/j.1360-0443.1990.tb01624.x. PMID 2285838
- [Background] Jonas DE, Amick HR, Feltner C, Bobashev G, Thomas K, Wines R, Kim MM, Shanahan E, Gass CE, Rowe CJ, Garbutt JC. Pharmacotherapy for adults with alcohol use disorders in outpatient settings: a systematic review and meta-analysis. JAMA. 2014 May 14;311(18):1889-900. doi: 10.1001/jama.2014.3628. PMID 24825644
- [Background] Kampman KM, Volpicelli JR, McGinnis DE, Alterman AI, Weinrieb RM, D'Angelo L, Epperson LE. Reliability and validity of the Cocaine Selective Severity Assessment. Addict Behav. 1998 Jul-Aug;23(4):449-61. doi: 10.1016/s0306-4603(98)00011-2. PMID 9698974
- [Background] Kendler KS, Ohlsson H, Maes HH, Sundquist K, Lichtenstein P, Sundquist J. A population-based Swedish Twin and Sibling Study of cannabis, stimulant and sedative abuse in men. Drug Alcohol Depend. 2015 Apr 1;149:49-54. doi: 10.1016/j.drugalcdep.2015.01.016. Epub 2015 Jan 28. PMID 25660314
- [Background] Kenward MG. Selection models for repeated measurements with non-random dropout: an illustration of sensitivity. Stat Med. 1998 Dec 15;17(23):2723-32. doi: 10.1002/(sici)1097-0258(19981215)17:233.0.co;2-5. PMID 9881418
- [Background] Kessler F, Cacciola J, Alterman A, Faller S, Souza-Formigoni ML, Cruz MS, Brasiliano S, Pechansky F. Psychometric properties of the sixth version of the Addiction Severity Index (ASI-6) in Brazil. Braz J Psychiatry. 2012 Mar;34(1):24-33. doi: 10.1590/s1516-44462012000100006. PMID 22392385
- [Background] Laird NM. Missing data in longitudinal studies. Stat Med. 1988 Jan-Feb;7(1-2):305-15. doi: 10.1002/sim.4780070131. PMID 3353609
- [Background] LaRowe SD, Mardikian P, Malcolm R, Myrick H, Kalivas P, McFarland K, Saladin M, McRae A, Brady K. Safety and tolerability of N-acetylcysteine in cocaine-dependent individuals. Am J Addict. 2006 Jan-Feb;15(1):105-10. doi: 10.1080/10550490500419169. PMID 16449100
- [Background] LaRowe SD, Myrick H, Hedden S, Mardikian P, Saladin M, McRae A, Brady K, Kalivas PW, Malcolm R. Is cocaine desire reduced by N-acetylcysteine? Am J Psychiatry. 2007 Jul;164(7):1115-7. doi: 10.1176/ajp.2007.164.7.1115. PMID 17606664
- [Background] Lussier JP, Heil SH, Mongeon JA, Badger GJ, Higgins ST. A meta-analysis of voucher-based reinforcement therapy for substance use disorders. Addiction. 2006 Feb;101(2):192-203. doi: 10.1111/j.1360-0443.2006.01311.x. PMID 16445548
- [Background] Lynskey MT, Agrawal A, Henders A, Nelson EC, Madden PA, Martin NG. An Australian twin study of cannabis and other illicit drug use and misuse, and other psychopathology. Twin Res Hum Genet. 2012 Oct;15(5):631-41. doi: 10.1017/thg.2012.41. Epub 2012 Jul 9. PMID 22874079
- [Background] Mardikian PN, LaRowe SD, Hedden S, Kalivas PW, Malcolm RJ. An open-label trial of N-acetylcysteine for the treatment of cocaine dependence: a pilot study. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Mar 30;31(2):389-94. doi: 10.1016/j.pnpbp.2006.10.001. Epub 2006 Nov 17. PMID 17113207
- [Background] McGinty JF, Mendelson JE. Is brain-derived neurotrophic factor a selective biomarker that predicts cocaine relapse outcomes? Biol Psychiatry. 2011 Oct 15;70(8):700-701. doi: 10.1016/j.biopsych.2011.08.017. No abstract available. PMID 21967984
- [Background] McGinty JF, Whitfield TW Jr, Berglind WJ. Brain-derived neurotrophic factor and cocaine addiction. Brain Res. 2010 Feb 16;1314:183-93. doi: 10.1016/j.brainres.2009.08.078. Epub 2009 Sep 2. PMID 19732758
- [Background] McLellan AT, Alterman AI, Cacciola J, Metzger D, O'Brien CP. A new measure of substance abuse treatment. Initial studies of the treatment services review. J Nerv Ment Dis. 1992 Feb;180(2):101-10. doi: 10.1097/00005053-199202000-00007. PMID 1737971
- [Background] McLellan AT, Kushner H, Metzger D, Peters R, Smith I, Grissom G, Pettinati H, Argeriou M. The Fifth Edition of the Addiction Severity Index. J Subst Abuse Treat. 1992;9(3):199-213. doi: 10.1016/0740-5472(92)90062-s. PMID 1334156
- [Background] Nestler EJ. From neurobiology to treatment: progress against addiction. Nat Neurosci. 2002 Nov;5 Suppl:1076-9. doi: 10.1038/nn945. PMID 12403990
- [Background] Nestler EJ. The neurobiology of cocaine addiction. Sci Pract Perspect. 2005 Dec;3(1):4-10. doi: 10.1151/spp05314. PMID 18552739
- [Background] Olive MF, Cleva RM, Kalivas PW, Malcolm RJ. Glutamatergic medications for the treatment of drug and behavioral addictions. Pharmacol Biochem Behav. 2012 Feb;100(4):801-10. doi: 10.1016/j.pbb.2011.04.015. Epub 2011 Apr 22. PMID 21536062
- [Background] de Lima Osorio F, Crippa JA, Loureiro SR. Further psychometric study of the Beck Anxiety Inventory including factorial analysis and social anxiety disorder screening. Int J Psychiatry Clin Pract. 2011 Nov;15(4):255-62. doi: 10.3109/13651501.2011.605955. PMID 22121998
- [Background] Patriquin MA, Bauer IE, Soares JC, Graham DP, Nielsen DA. Addiction pharmacogenetics: a systematic review of the genetic variation of the dopaminergic system. Psychiatr Genet. 2015 Oct;25(5):181-93. doi: 10.1097/YPG.0000000000000095. PMID 26146874
- [Background] Pavanello S, Hoxha M, Dioni L, Bertazzi PA, Snenghi R, Nalesso A, Ferrara SD, Montisci M, Baccarelli A. Shortened telomeres in individuals with abuse in alcohol consumption. Int J Cancer. 2011 Aug 15;129(4):983-92. doi: 10.1002/ijc.25999. Epub 2011 Apr 25. PMID 21351086
- [Background] Prendergast M, Podus D, Finney J, Greenwell L, Roll J. Contingency management for treatment of substance use disorders: a meta-analysis. Addiction. 2006 Nov;101(11):1546-60. doi: 10.1111/j.1360-0443.2006.01581.x. PMID 17034434
- [Background] Rabkin JG, Markowitz JS, Ocepek-Welikson K, Wager SS. General versus systematic inquiry about emergent clinical events with SAFTEE: implications for clinical research. J Clin Psychopharmacol. 1992 Feb;12(1):3-10. doi: 10.1097/00001573-199202000-00002. PMID 1552037
- [Background] Rosa AR, Sanchez-Moreno J, Martinez-Aran A, Salamero M, Torrent C, Reinares M, Comes M, Colom F, Van Riel W, Ayuso-Mateos JL, Kapczinski F, Vieta E. Validity and reliability of the Functioning Assessment Short Test (FAST) in bipolar disorder. Clin Pract Epidemiol Ment Health. 2007 Jun 7;3:5. doi: 10.1186/1745-0179-3-5. PMID 17555558
- [Background] Sansone RA, Sansone LA. Getting a Knack for NAC: N-Acetyl-Cysteine. Innov Clin Neurosci. 2011 Jan;8(1):10-4. PMID 21311702
- [Background] Santos Cruz M, Andrade T, Bastos FI, Leal E, Bertoni N, Villar LM, Tiesmaki M, Fischer B. Key drug use, health and socio-economic characteristics of young crack users in two Brazilian cities. Int J Drug Policy. 2013 Sep;24(5):432-8. doi: 10.1016/j.drugpo.2013.03.012. Epub 2013 Apr 28. PMID 23632130
- [Background] Schmaal L, Berk L, Hulstijn KP, Cousijn J, Wiers RW, van den Brink W. Efficacy of N-acetylcysteine in the treatment of nicotine dependence: a double-blind placebo-controlled pilot study. Eur Addict Res. 2011;17(4):211-6. doi: 10.1159/000327682. Epub 2011 May 24. PMID 21606648
- [Background] Schmaal L, Veltman DJ, Nederveen A, van den Brink W, Goudriaan AE. N-acetylcysteine normalizes glutamate levels in cocaine-dependent patients: a randomized crossover magnetic resonance spectroscopy study. Neuropsychopharmacology. 2012 Aug;37(9):2143-52. doi: 10.1038/npp.2012.66. Epub 2012 May 2. PMID 22549117
- [Background] Schneider R Jr, Santos CF, Clarimundo V, Dalmaz C, Elisabetsky E, Gomez R. N-acetylcysteine prevents behavioral and biochemical changes induced by alcohol cessation in rats. Alcohol. 2015 May;49(3):259-63. doi: 10.1016/j.alcohol.2015.01.009. Epub 2015 Feb 13. PMID 25771148
- [Background] Shen Q, Zhao X, Yu L, Zhang Z, Zhou D, Kan M, Zhang D, Cao L, Xing Q, Yang Y, Xu H, He L, Liu Y. Association of leukocyte telomere length with type 2 diabetes in mainland Chinese populations. J Clin Endocrinol Metab. 2012 Apr;97(4):1371-4. doi: 10.1210/jc.2011-1562. Epub 2012 Feb 8. PMID 22319045
- [Background] Sinha R. New findings on biological factors predicting addiction relapse vulnerability. Curr Psychiatry Rep. 2011 Oct;13(5):398-405. doi: 10.1007/s11920-011-0224-0. PMID 21792580
- [Background] Skinner MD, Lahmek P, Pham H, Aubin HJ. Disulfiram efficacy in the treatment of alcohol dependence: a meta-analysis. PLoS One. 2014 Feb 10;9(2):e87366. doi: 10.1371/journal.pone.0087366. eCollection 2014. PMID 24520330
- [Background] Sordi AO, Pechansky F, Kessler FH, Kapczinski F, Pfaffenseller B, Gubert C, de Aguiar BW, de Magalhaes Narvaez JC, Ornell F, von Diemen L. Oxidative stress and BDNF as possible markers for the severity of crack cocaine use in early withdrawal. Psychopharmacology (Berl). 2014 Oct;231(20):4031-9. doi: 10.1007/s00213-014-3542-1. Epub 2014 Mar 28. PMID 24676990
- [Background] Spencer RL, Hutchison KE. Alcohol, aging, and the stress response. Alcohol Res Health. 1999;23(4):272-83. PMID 10890824
- [Background] Sullivan JT, Sykora K, Schneiderman J, Naranjo CA, Sellers EM. Assessment of alcohol withdrawal: the revised clinical institute withdrawal assessment for alcohol scale (CIWA-Ar). Br J Addict. 1989 Nov;84(11):1353-7. doi: 10.1111/j.1360-0443.1989.tb00737.x. PMID 2597811
- [Background] Urbanska EM, Czuczwar SJ, Kleinrok Z, Turski WA. Excitatory amino acids in epilepsy. Restor Neurol Neurosci. 1998;13(1-2):25-39. PMID 12671285
- [Background] Verdejo-Garcia A, Perez-Garcia M. Profile of executive deficits in cocaine and heroin polysubstance users: common and differential effects on separate executive components. Psychopharmacology (Berl). 2007 Mar;190(4):517-30. doi: 10.1007/s00213-006-0632-8. Epub 2006 Nov 29. PMID 17136401
- [Background] Volkow ND, Koob G, Baler R. Biomarkers in substance use disorders. ACS Chem Neurosci. 2015 Apr 15;6(4):522-5. doi: 10.1021/acschemneuro.5b00067. Epub 2015 Mar 18. PMID 25734247
- [Background] von Diemen L, Kapczinski F, Sordi AO, de Magalhaes Narvaez JC, Guimaraes LS, Kessler FH, Pfaffenseller B, de Aguiar BW, de Moura Gubert C, Pechansky F. Increase in brain-derived neurotrophic factor expression in early crack cocaine withdrawal. Int J Neuropsychopharmacol. 2014 Jan;17(1):33-40. doi: 10.1017/S146114571300103X. Epub 2013 Sep 26. PMID 24067327
- [Background] Walker J, Winhusen T, Storkson JM, Lewis D, Pariza MW, Somoza E, Somoza V. Total antioxidant capacity is significantly lower in cocaine-dependent and methamphetamine-dependent patients relative to normal controls: results from a preliminary study. Hum Psychopharmacol. 2014 Nov;29(6):537-43. doi: 10.1002/hup.2430. PMID 25087849
- [Background] Wei LJ, Lachin JM. Properties of the urn randomization in clinical trials. Control Clin Trials. 1988 Dec;9(4):345-64. doi: 10.1016/0197-2456(88)90048-7. PMID 3203525
- [Background] Wu Y, Pan X, Zhang S, Wang W, Cai M, Li Y, Yang F, Guo H. Protective effect of corn peptides against alcoholic liver injury in men with chronic alcohol consumption: a randomized double-blind placebo-controlled study. Lipids Health Dis. 2014 Dec 13;13:192. doi: 10.1186/1476-511X-13-192. PMID 25494594
- [Background] Yang Z, Ye J, Li C, Zhou D, Shen Q, Wu J, Cao L, Wang T, Cui D, He S, Qi G, He L, Liu Y. Drug addiction is associated with leukocyte telomere length. Sci Rep. 2013;3:1542. doi: 10.1038/srep01542. PMID 23528991
- [Background] Zaparte A, Viola TW, Grassi-Oliveira R, da Silva Morrone M, Moreira JC, Bauer ME. Early abstinence of crack-cocaine is effective to attenuate oxidative stress and to improve antioxidant defences. Psychopharmacology (Berl). 2015 Apr;232(8):1405-13. doi: 10.1007/s00213-014-3779-8. Epub 2014 Oct 23. PMID 25338778
- [Background] Zhou W, Kalivas PW. N-acetylcysteine reduces extinction responding and induces enduring reductions in cue- and heroin-induced drug-seeking. Biol Psychiatry. 2008 Feb 1;63(3):338-40. doi: 10.1016/j.biopsych.2007.06.008. Epub 2007 Aug 24. PMID 17719565